CLINICAL TRIAL: NCT02338739
Title: An Adaptive Strategy for Preventing and Treating Lapses of Retention in Adult HIV Care (AdaPT-R)
Brief Title: An Adaptive Strategy for Preventing and Treating Lapses of Retention in Adult HIV Care (AdaPT-R) in Nyanza, Kenya
Acronym: AdaPT-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Kenya Medical Research Institute (Other); University of Washington (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01MH104123-01 (NIH); 1R01MH104123-01 (NIH)
Record Dates: First submitted 2014-12-11; First posted 2015-01-14 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: Retention; Lost to follow up; Adaptive strategies; Dynamic regime; Sequentially randomized trial; Sequential multiple assignment randomized trial; Engagement in care; Kenya
MeSH Terms: interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (15):
- REC; Outreach if Failure (Active Comparator)
  Interventions: Behavioral: REC; Outreach if Failure
- REC; SMS + Voucher if Failure (Active Comparator)
  Interventions: Behavioral: REC; SMS + Voucher if Failure
- REC; Navigator if Failure (Active Comparator)
  Interventions: Behavioral: REC; Navigator if Failure
- SMS; Outreach if Failure (Active Comparator)
  Interventions: Behavioral: SMS; Outreach if Failure
- SMS; Outreach if Failure; Stop SMS if Success (Active Comparator)
  Interventions: Behavioral: SMS; Outreach if Failure; Stop SMS if Success
- SMS; SMS+Voucher if Failure (Active Comparator)
  Interventions: Behavioral: SMS; SMS+Voucher if Failure
- SMS; SMS+Voucher if Failure; Stop SMS if Success (Active Comparator)
  Interventions: Behavioral: SMS; SMS+Voucher if Failure; Stop SMS if Success
- SMS; Navigator if Failure (Active Comparator)
  Interventions: Behavioral: SMS; Navigator if Failure
- SMS; Navigator if Failure; Stop SMS if Success (Active Comparator)
  Interventions: Behavioral: SMS; Navigator if Failure; Stop SMS if Success
- Voucher; Outreach if Failure (Active Comparator)
  Interventions: Behavioral: Voucher; Outreach if Failure
- Voucher; Outreach if Failure; Stop Voucher if Success (Active Comparator)
  Interventions: Behavioral: Voucher; Outreach if Failure; Stop Voucher if Success
- Voucher; SMS+Voucher if Failure (Active Comparator)
  Interventions: Behavioral: Voucher; SMS+Voucher if Failure
- Voucher; SMS+Voucher if Failure; Stop Voucher if Success (Active Comparator)
  Interventions: Behavioral: Voucher; SMS+Voucher if Failure; Stop Voucher if Success
- Voucher; Navigator if Failure (Active Comparator)
  Interventions: Behavioral: Voucher; Navigator if Failure
- Voucher; Navigator if Failure; Stop Voucher if Success (Active Comparator)
  Interventions: Behavioral: Voucher; Navigator if Failure; Stop Voucher if Success

INTERVENTIONS:
Behavioral: REC; Outreach if Failure — Routine education and counseling (REC) services, delivered per Kenya Ministry of Health Guidelines; followed by standard of care (SOC) outreach to encourage return to clinic for patients 14 days late for a scheduled visit in year 1.
  Arms: REC; Outreach if Failure
Behavioral: REC; SMS + Voucher if Failure — Routine education and counseling services, delivered per Kenya Ministry of Health (MOH) Guidelines; followed by SMS text messages for patients and reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients 14 days late for a scheduled visit in year 1.
  Arms: REC; SMS + Voucher if Failure
Behavioral: REC; Navigator if Failure — REC services, delivered per Kenya MOH Guidelines; followed by Peer Navigator (tailored outreach and support) for patients 14 days late for a scheduled visit
  Arms: REC; Navigator if Failure
Behavioral: SMS; Outreach if Failure — SMS text messages for patients; followed by SOC outreach for patients 14 days late for a scheduled visit
  Arms: SMS; Outreach if Failure
Behavioral: SMS; Outreach if Failure; Stop SMS if Success — SMS text messages for patients, followed by SOC outreach for patients 14 days late for a scheduled visit, and discontinuation of SMS text messages if never 14 days late
  Arms: SMS; Outreach if Failure; Stop SMS if Success
Behavioral: SMS; SMS+Voucher if Failure — SMS text messages for patients, followed by reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients 14 days late for a scheduled visit in year 1.
  Arms: SMS; SMS+Voucher if Failure
Behavioral: SMS; SMS+Voucher if Failure; Stop SMS if Success — SMS text messages for patients, followed by reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients 14 days late for a scheduled visit in year 1, and discontinuation of SMS text messages if never 14 days late
  Arms: SMS; SMS+Voucher if Failure; Stop SMS if Success
Behavioral: SMS; Navigator if Failure — SMS text messages for patents, followed by Peer Navigator (tailored outreach and support) for patients 14 days late for a scheduled visit
  Arms: SMS; Navigator if Failure
Behavioral: SMS; Navigator if Failure; Stop SMS if Success — SMS text messages for patents, followed by Peer Navigator (tailored outreach and support) for patients 14 days late for a scheduled visit, and discontinuation of SMS text messages if never 14 days late
  Arms: SMS; Navigator if Failure; Stop SMS if Success
Behavioral: Voucher; Outreach if Failure — Reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients, followed by SOC outreach for patients 14 days late for a scheduled visit
  Arms: Voucher; Outreach if Failure
Behavioral: Voucher; Outreach if Failure; Stop Voucher if Success — Reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients, followed by SOC outreach for patients 14 days late for a scheduled visit, and discontinuation of voucher for patients if never 14 days late
  Arms: Voucher; Outreach if Failure; Stop Voucher if Success
Behavioral: Voucher; SMS+Voucher if Failure — Reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients, followed by SMS text message and reimbursement (KSH 400) for transport to the clinic for patients 14 days late for a scheduled visit
  Arms: Voucher; SMS+Voucher if Failure
Behavioral: Voucher; SMS+Voucher if Failure; Stop Voucher if Success — Reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients, followed by SMS text message and reimbursement (KSH 400) for transport to the clinic for patients 14 days late for a scheduled visit, and discontinuation of voucher for patients if never 14 days late
  Arms: Voucher; SMS+Voucher if Failure; Stop Voucher if Success
Behavioral: Voucher; Navigator if Failure — Reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients, followed by Peer Navigator (tailored outreach and support) for patients 14 days late for a scheduled visit
  Arms: Voucher; Navigator if Failure
Behavioral: Voucher; Navigator if Failure; Stop Voucher if Success — Reimbursement at a fixed amount (KSH 400) for transport to the clinic for patients, followed by Peer Navigator (tailored outreach and support) for patients 14 days late for a scheduled visit, and discontinuation of voucher for patients if never 14 days late
  Arms: Voucher; Navigator if Failure; Stop Voucher if Success

SUMMARY:
Retaining HIV-infected patients in care is critical, but loss to follow-up after enrolment often reaches 20%-40% by two years, placing millions of patients at risk of poor outcomes. A strategy to optimize retention within resource constraints is urgently needed. Sequential adaptive strategies - a novel class of public health approaches - may offer a solution. A candidate sequential adaptive strategy would start with a less expensive intervention (e.g., SMS) in all patients and then apply a more costly and intensive one (e.g., navigator) only to patients who show early signs of poor retention. This study involves a sequential multiple assignment randomized trial to evaluate a family of such strategies. the investigators will randomize 1,800 adults newly initiating antiretroviral treatment (ART) at 4 HIV clinics in the Nyanza region of Kenya to (1) standard of care routine education and counselling (REC), (2) SMS text messages, or (3) transport vouchers. Patients with early signs of weakening retention (defined as the first time a patient is 14 days late for an appointment) will be re-randomized to (1) a single episode of outreach (standard of care), (2) SMS combined with vouchers, or (3) a peer navigator. Patients not successfully contacted by 28 days after missed visit (and not verified to have left the area or transferred to another clinic) will also be rerandomized to of one the same three re-engagement interventions. Individuals randomized at first stage to SMS or voucher that do not miss a visit by at least 14 days in the first 12 months of follow up will be re-randomized at 12 months to stop first stage intervention or continue with that same intervention to 24 months. The investigators primary objective is to assess the comparative effectiveness of sequenced intervention strategies to prevent initial lapses in retention and to treat those that occur. The investigators primary endpoint is fraction of time retained in care two years after enrolment. In addition, the investigators will assess the comparative effectiveness of first-stage strategies (REC, SMS, voucher) to prevent lapses in retention, and the comparative effectiveness of second stage strategies (outreach, SMS + voucher, navigator) to re-engage patients after initial lapse. This study will also compare outcomes among patients who continue versus discontinue the SMS and voucher interventions, including a small complementarity component utilizing qualitative methods to examine the voucher approach and the effects of discontinuing this approach after success among a subset of participants. At study conclusion the investigators output will be a menu of adaptive strategies for retention, accompanied by estimates of cost and effectiveness, which policy makers in different settings can use to advance the impact of HIV care and treatment programs in Africa.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* 18 years old
* Planning to remain in the study area (Nyanza region) for the duration of the study, capable of informed consent
* Newly initiating ART (within past 90 days)
* Access to a cell phone
* Ability to read or be read SMS messages
* And willingness to be contacted by clinic upon missed appointment.

Exclusion Criteria:

* Plans to move out of Nyanza region or acutely ill and requiring hospitalization.
* Hospitalized patients who later recover will be eligible for enrolment at the first post-hospitalization clinic visit during which eligibility criteria are met.
* No access to a cell phone.
* Involvement in studies with the potential to influence retention behaviors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1816 (Actual)
Dates: Start 2015-03; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Retention | Up to two years after enrollment
  Fraction of time in care

SECONDARY OUTCOMES:
Alive with suppressed HIV RNA level (<400 copies/ml) | Two years after study enrollment
  Number of subjects alive with suppressed HIV RNA levels (<400 copies/ml)
Time from second randomization to return to clinic after initial retention lapse | Up to two years after enrollment
  Time from second randomization to re-engagement; re-engagement is defined as first visit back to clinic
Mean visit adherence (% visits made) | Two years after study enrollment
  Proportion of kept scheduled appointments (range=0-100%), with kept visits being those attended by the patient and with the denominator excluding canceled visits
Retention | Two years after enrollment
  Fraction of time in care
Fraction on-time pharmacy pick-ups for antiretroviral drugs | Two years after enrollment
  Proportion of prescriptions filled and picked up by participants to prescriptions written
Cost effectiveness | After two years of enrollment
  Cost per failure (virological failure (HIV RNA>=400 copies/ml) or death averted
Patient-reported barriers to engagement | At years one and two after study enrollment
  Self-reported by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elvin Geng, MD, Principal Investigator — University of California, San Francisco; Maya Petersen, MD, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- Kenya Medical Research Institute, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Geng EH, Odeny TA, Montoya LM, Iguna S, Kulzer JL, Adhiambo HF, Eshun-Wilson I, Akama E, Nyandieka E, Guze MA, Shade S, Packel L, Fox B, Camlin C, Thirumurthy H, Lyons C, Bukusi EA, Petersen ML. Adaptive Strategies for Retention in Care among Persons Living with HIV. NEJM Evid. 2023 Apr;2(4):10.1056/evidoa2200076. doi: 10.1056/evidoa2200076. Epub 2023 Mar 28. PMID 38143482